CLINICAL TRIAL: NCT05656547
Title: Anesthetic Sparing Effects of Dexmedetomidine During Craniotomy: a Retrospective Propensity Score Matching Comparison Between Encephalographic Spectrogram-guided and Processes Encephalographic Index-guided Protocol
Brief Title: EEG DSA-guided Intravenous Anesthesia Using Dexmedetomidine and Propofol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202211078RINC
Record Dates: First submitted 2022-12-11; First posted 2022-12-19 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Brain Surgery
Keywords: electroencephalogram; dexmedetomidine; total intravenous anesthesia; craniotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Encephalographic spectrogram group: The dexmedetomidine and propofol infusions were titrated to maintain robust alpha power in the encephalographic spectrogram
- Encephalographic index group: The dexmedetomidine and propofol infusions were titrated to maintain the bispectral index score between 40 and 60.

SUMMARY:
Investigators conduct this retrospective analysis to test this hypothesis that the EEG spectrogram guided general anesthesia with dexmedetomidine co-administration with propofol may significantly reduce the propofol consumption during craniotomy and to investigate potential benefits on postoperative outcomes.

DETAILED DESCRIPTION:
The bispectral index (BIS), is widely applied to maintain anesthetic depth. However, this processed EEG index may be ambiguous when dexmedetomidine is administrated. Because each anesthetic produces distinct brain states that are readily visible in the EEG spectrogram which can be easily interpreted by anesthesiologists, the EEG spectrogram-guided anesthesia is theoretically beneficial to avoid unnecessary anesthetic exposure when dexmedetomidine is co-administrated but this remains not yet clarified. Recently, the investigators reported a randomized controlled trial which revealed that co-administration of dexmedetomidine with propofol by using the BIS score guidance, is associated with profound propofol sparing effects and more favorable postoperative neurological outcomes (Eur J Anaesthesiol . 2021 Dec 1;38(12):1262-1271.). Based on the advance of knowledge of EEG spectrogram, the investigators have transited our practice based on the EEG spectrogram guidance. In this study, the investigators analyze the influence of EEG spectrogram guidance on the propofol sparing effect and the postoperative profile in comparison to patients of our previous BIS-guided protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective craniotomy for brain tumor resection, aneurysm clipping, an intracranial bypass procedure, or microvascular decompression
* age between 20 to 80 yr

Exclusion Criteria:

* Fever, elevated white blood cell or C-reactive protein
* Impaired liver function, eg. AST or ALT >100; liver cirrhosis > Child B class
* Impaired renal function, cGFR< 60 ml/min/1.73 m2
* Cardiac dysfunction, such as heart failure > NYHA class II

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective craniotomy for brain tumor resection, aneurysm clipping, an intracranial bypass procedure, or microvascular decompression.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-01-25 (Estimated); Study Completion 2023-02-25 (Estimated)

PRIMARY OUTCOMES:
Propofol dose requirement | 4-6 hours
  Intraoperative propofol consumption

SECONDARY OUTCOMES:
Postoperative delirium | During hospital stay, estimated 7-10 days
  Postoperative delirium diagnosed using the Intensive Care Delirium Screening Checklist (ICDSC) criteria
Postoperative Barthel index change | During hospital stay, estimated 7-10 days
  Barthel index changes between the states of admission and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan